CLINICAL TRIAL: NCT06688396
Title: Dilated Cardiomyopathy Detection Using Artificial Intelligence and Screening With Mobile Technology
Brief Title: Dilated Cardiomyopathy Detection Using AI and Screening With Mobile Technology (DCM-DETECT)
Acronym: DCM-DETECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lancaster General Hospital (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 855484
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Dilated Cardiomyopathy; Heart Failure; Heart Disease
Keywords: Dilated Cardiomyopathy; Heart Failure; Heart Disease
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- DCM Screening (Experimental): Participants (probands) with dilated cardiomyopathy (DCM) will invite their first-degree relatives (FDR) to participate in DCM screening to examine the impact of an "Artificial Intelligent" (AI) enhanced 6lead (6L) mobile electrocardiogram (EKG) in encouraging FDR of probands with a DCM to obtain appropriate cardiac screening.
  Interventions: Device: Mobile 6L AI-EKG Screening

INTERVENTIONS:
Device: Mobile 6L AI-EKG Screening — Participants (probands) with DCM will invite their first-degree relatives to undergo DCM screening procedures.
  Probands and first-degree relatives will complete a mobile 6L AI-EKG which will be transmitted to a mobile app and interpreted by the AI-EKG algorithm. Results will be shared electronically or verbally to the participant.
  If available, the probands clinical 12L EKGs will be obtained if recorded within 30 days of their Kardia 6L recording.
  All participating FDR will be encouraged to pursue cardiac screening per ACC/AHA recommendations. Study staff will obtain echocardiogram results up to 6 months of participant enrollment.

SUMMARY:
This is a prospective, single-arm clinical trial in which participants with dilated cardiomyopathy will invite their first degree relatives to undergo mobile cardiac, electrocardiogram screening.

DETAILED DESCRIPTION:
The purpose of this study is to examine the impact of an "Artificial Intelligent" (AI) enhanced 6Lead (6L) mobile electrocardiogram (EKG) in encouraging first degree relatives (FDR) of probands with a dilated cardiomyopathy (DCM) to obtain appropriate cardiac screening.

The AI enhanced EKG (AI-EKG) will be acquired using the AliveCor KardiaMobile 6L system which allows the generation of prediction probabilities for reduced left ventricular function (LVEF). The AliveCor KardiaMobile 6L device is an FDA approved handheld smart device that records an EKG in 30 seconds to 5-minute increments. The device is an ambulatory wireless device that connects to a smartphone and is easy to use. The EKG signal is communicated wirelessly via Bluetooth to a mobile computing platform (MCP) which can be a smartphone or tablet. The MCP will be running either the KardiaRx mobile application if the participant is remote, or the KardiaStation App if the participation is on sight at either the Lancaster General Hospital (LGH) campus or the Central Pennsylvania Clinic (CPC) location. The 6L EKG is transmitted following processing by the Kardia Apps. The results of the EKG tracings recorded by the AliveCor devices will not be entered into the electronic medical record or used to guide clinical care. The EKG data from the recordings identified only by the connection code will be uploaded to the AliveCor cloud for proprietary AI analysis designed to detect impaired LVEF. This AI software for LVEF analysis is FDA approved.

All participating FDR will be encouraged to pursue cardiac screening per American College of Cardiology/American Heart Association (ACC/AHA) recommendations.

If available, the probands clinical 12Lead (12L) EKGs will be obtained if recorded within 30 days of their Kardia 6L recording. The concordance of the algorithm results applied to the Kardia 6L data with the 12L FDA approved LVEF algorithm results will be assessed.

ELIGIBILITY:
Inclusion Criteria (Proband)

* Male or female age ≥ 18 years
* Confirmed diagnosis of non-ischemic DCM determined at the discretion of the treating physician and defined as LVEF ≤ 45% at any time during the clinical course of the patient
* Must have at least one living adult FDR
* Able to provide informed consent

Inclusion Criteria (FDR)

* Male or female age ≥ 18 years who are first-degree relatives of patients with DCM
* Proband has provided informed consent
* FDR able to provide informed verbal consent
* Access to a smartphone or digital tablet with cellular data or Wi-Fi access

Exclusion Criteria (Proband)

* DCM attributed to any other secondary form of cardiomyopathy per the investigator's determination
* Proband has previously informed FDR to undergo cardiac screening
* Ischemic cause of reduced LVEF

  * evidence of myocardial infarction, inducible ischemia or chest pain on stress testing in absence of coronary angiogram to rule out ischemic disease
  * history of acute coronary syndromes (STEMI (ST-Elevation Myocardial Infarction), NSTEMI (Non-ST-Elevation Myocardial Infarction) or unstable angina) revascularization or ≥75% stenosis of either left main or Left Anterior Descending (LAD) or ≥75% stenosis of 2 major epicardial vessels on angiogram
* Moderate or greater primary valvular abnormality not due to underlying cardiomyopathy
* Congenital structural heart disease
* Severe and untreated or untreatable hypertension
* Cardiomyopathy due to acute or reversible conditions; examples include tachyarrhythmias, thyroid disorders, iron overload
* Any secondary cause of reduced LVEF such as pregnancy, myocarditis, amyloidosis, sarcoidosis, exposure to toxins including alcohol, substance abuse or chemotherapeutic drug
* (CPC Participants only) Home address outside of traveling range

Exclusion Criteria (FDR)

* Previously informed about cardiac screening or has completed cardiac screening by transthoracic echocardiogram (TTE)
* Previously diagnosed with reduced LVEF
* (CPC Participants only) Home address outside of traveling range

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
This study's primary endpoint is to assess the feasibility of performing AI-EKG test and the subsequent uptake of cardiac screening in FDR of DCM patients. | Assessed for a minimum of 3 months post enrollment up to 6 months post enrollment.
  The number of consented FDR who successfully undergo AI-EKG and subsequent recommended cardiac follow up.

SECONDARY OUTCOMES:
Positive AI-EKG screens among FDR of DCM probands (LVEF ≤ 45%)/total population of the FDR of DCM probands undergoing AI-EKG. | Assessed at time of EKG results. About 2 weeks post collection.

OTHER OUTCOMES:
Responses to decliner survey questions addressing barriers to adoption of AI technology, variables that contribute to the reluctance to participate, and logistical barriers to research. surveys. | Assessed at time of decline and survey completion, about 30 minutes.
Positive cardiac screening procedures /total number of FDR undergoing cardiac screening procedures | Assessed at 3 months post enrollment check-in or 6 months post enrollment check-in if not completed by 3 months.
Comparison of AI EKG reduced LVEF algorithm results between 6L Kardia EKG and 12L AI EKG, if available, in DCM probands. | Assessed during data analysis, 2 years after study start.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Small, MD, Principal Investigator — Penn Medicine / Lancaster General Hospital
Locations (1):
- Lancaster General Hospital, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Proposed Regulatory Framework for Modifications to Artificial Intelligence/Machine Learning (AI/ML)-Based Software as a Medical Device (SaMD). — https://www.fda.gov/files/medical%20devices/published/US-FDA-Artificial-Intelligence-and-Machine-Learning-Discussion-Paper.pdf
- See also: Investigational Device Exemptions — https://www.ecfr.gov/current/title-21/chapter-1/subchapter-H/part-812
- See also: Information Sheet Guidance for IRBs, Clinical Investigators, and Sponsors — https://www.fda.gov/media/75459/download